CLINICAL TRIAL: NCT03099356
Title: An Open Label Phase II Trial Evaluating the Efficacy of Cyclophosphamide and Sirolimus for the Treatment of Metastatic, RAI-refractory, Differentiated Thyroid Cancer
Brief Title: Cyclophosphamide and Sirolimus for the Treatment of Metastatic, RAI-refractory, Differentiated Thyroid Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2017.013; HUM00126559 (Other: University of Michigan)
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Cyclophosphamide; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cyclophosphamide and Sirolimus (Experimental): Sirolimus 4 mg, PO, days 1-28 as well as Cyclophosphamide 100 mg, PO, days 1-5 and 15-19
  Interventions: Drug: Cyclophosphamide; Drug: Sirolimus

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide 100 mg, PO, days 1-5 and 15-19
Drug: Sirolimus — Sirolimus 4 mg, PO, days 1-28

SUMMARY:
This study will be a non-randomized pilot trial using Cyclophosphamide and Sirolimus for the treatment of metastatic differentiated thyroid cancer. Patients will be treated with Sirolimus 4 mg, PO, days 1-28 as well as Cyclophosphamide 100 mg, PO, days 1-5 and 15-19. Cycle length will be 28 days. Patients will be monitored closely for toxicity and undergo imaging to evaluate efficacy once every 2 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented differentiated thyroid cancer with or without metastases, not amenable to curative treatment; or the patient has documented refusal of curative treatment
* Measurable disease (>10 mm) and have progression of disease based on RECIST criteria. Previously irradiated tumor lesions are not considered measurable unless they have progressed since radiation.
* Previous failure of Iodine-131 (131I) therapy or not candidates to receive 131I as assessed by treating physician.
* Age ≥ 18 years
* ECOG (Eastern Cooperative Oncology Group) performance status 0-2
* Life expectance of ≥ 12 weeks
* 131I therapy not allowed within 24 weeks before entry (4 weeks if negative post-treatment scan)
* Adequate organ and marrow function
* Women of childbearing potential must have a negative serum or urine pregnancy test within 3 days prior to treatment
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment
* Willingness and ability to comply with scheduled visits, treatment plans, including willingness to take study medication, laboratory tests, and other study procedures

Exclusion Criteria:

* Inability to obtain Foundation One testing on archival tissue, or, lack of previous Next Generation Sequencing
* Chemotherapy, tyrosine kinase inhibitor, or radiation therapy within 4 weeks
* Prior experimental therapy within 4 weeks of planned start of this trial
* 131I therapy within 24 weeks before entry (4 weeks if negative post-treatment scan)
* Previous treatment with an mTOR inhibitor
* Patients who are currently receiving treatment with strong inhibitors or inducers of CYP3A4 or P-glycoprotein that cannot be discontinued at least one week prior to the start of treatment with Cyclophosphamide and Sirolimus
* Impairment of GI (gastrointestinal) function or GI disease that may significantly alter the absorption of study medications (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection) including dependence on a G-Tube for administration of medications.
* A serious uncontrolled medical disorder or active infection that would impair their ability to receive study treatment
* Patients with known sensitivities to either cyclophosphamide and/or sirolimus
* Patients with known urinary outflow obstruction
* Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol
* Patients (male and female) having procreative potential who are not willing or not able to use adequate contraception or practicing abstinence
* Women who are pregnant or breast-feeding
* Patients residing in prison

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2017-04-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients that respond to treatment | Patients will be followed for response until progression or up to 2 Years
  The primary measure of efficacy will be the overall response rate (ORR) which is defined as those achieving either complete response (CR) or partial response (PR). Partial response is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions. Complete response is defined as Disappearance of all target lesions, determined by two separate observations conducted not less than 4 weeks apart (there can be no appearance of new lesions) and the disappearance of all non-target lesions and normalization of tumor marker level.

SECONDARY OUTCOMES:
The number of patients that experience toxicity | Patients are followed for toxicity up to 30 days after the last dose of study drug
  The number of patients that experience toxicity by type will be reported.
Median overall survival time | Patients will be followed until death or up to 2 years
  The median duration of time from start of treatment until death
Median progression free survival time | Patients will be followed for response until progression or up to 2 Years
  The median duration of time from start of treatment until progression. Progression is defined as at least a 20% increase in the sum of the LD (longest diameter) of target lesions, taking as reference the smallest sum LD recorded since the treatment started, or the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Swiecicki, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States